CLINICAL TRIAL: NCT05956119
Title: Analysis of the Effectiveness of Dry Needling for Improving Gait in the Patient With Multiple Sclerosis: a Randomized Single-blind Clinical Trial
Brief Title: Effectiveness of Dry Needling for Improving Gait in the Patient With Multiple Sclerosis
Acronym: DRYNEEDEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario de Canarias (Other)
Responsible Party: Principal Investigator, Alberto Javier Ormazábal, Principal Investigator, Hospital Universitario de Canarias
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CHUC_2023_40
Record Dates: First submitted 2023-07-11; First posted 2023-07-21 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Dry Needling; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dry needling (Experimental): The intervention group will have a single session of dry nedling application in the medial gastrocnemius + usual care (physiotherapy)
  Interventions: Device: dry needling + physiotherapy (standard/usual care)
- placebo (Sham Comparator): The control group will have a single session of sham dry nedling in the medial gastrocnemius + usual care (physiotherapy)
  Interventions: Other: sham dry needling + physiotherapy (standard/usual care)

INTERVENTIONS:
Device: dry needling + physiotherapy (standard/usual care) — same that arm descrption
  Arms: dry needling
Other: sham dry needling + physiotherapy (standard/usual care) — same that arm description
  Arms: placebo

SUMMARY:
Multiple sclerosis (MS) is a chronic, inflammatory, autoimmune disease characterized by the appearance of lesions, characterized by heterogeneity in its pathological, clinical and radiological presentation. It has a significant socioeconomic impact, affecting interpersonal relationships and causing a significant reduction in quality of life.

Patients with MS suffer from a series of symptoms (ocular, spasticity, cerebellar, sensory, fatigue, depression) that may be independent of the course of the disease and their management significantly influences quality of life and also requires multidisciplinary therapeutic measures.

Physiotherapy and occupational therapy techniques are essential to reduce spasticity and prevent complications derived from it. Amongst physiotherapy techniques, we can find minimally invasive techniques such as dry needling which uses a fine filiform needle to penetrate the skin and mechanically break the myofascial trigger points, charactewrized by abnomral/pathological electrical activity. There have been previous studies with dry needling in stroke patients which have shown improvements in gait, but its effectiveness in other populations such as multiple sclerosis is still unclear.

In addition, dry needling has proven to be a cost-effective treatment for spasticity in patients with chronic and subacute stroke and could be an alternative to other pharmacological treatments, although more studies are necessary to compare both the effectiveness and the cost-effectiveness .

Recent studies carried out in patients with multiple sclerosis suggest that dry needling can improve mobility and gait speed. The main objective of the study is to analyze the effect of the application of a single session of dry needling in the lower limbs on the gait of patients with multiple sclerosis.

A prospective randomized parallel group clinical trial with blinded outcome assessment will be conducted. Participants will be recruited from the Hospital Universitario de Canarias.

ELIGIBILITY:
Inclusion Criteria:

1. Having been diagnosed with Multiple Sclerosis in a period of more than two years before the study starts
2. Participate voluntarily and sign the informed consent.
3. Suffering from some type of hypertonia or spasticity in MMII that makes walking difficult, measured with Expanded Disability Status Scale>2 (Pyramidal section >2)
4. Age from 18 to 60 years old.
5. Not having phobia of needles.

Exclusion Criteria:

1. Not signing the informed consent.
2. Having a phobia of needles.
3. Presenting an outbreak at the start of the study or having presented any outbreak up to two months before the start of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Change in Timed 25-Foot Walk (T25FW) | inmediatly before intervention, inmediatly after intervention, a week after the intervention and a month after the intervention
  is a quantitative mobility and leg function performance test based on a timed 25-walk. This is considered the "gold standard" to assess gait speed in MS patients. The test measures the time in seconds that the patient needs to walk 25 feet (7.5 meters).

SECONDARY OUTCOMES:
Change in Multiple Sclerosis Walking Scale (MSWS-12) | inmediatly before intervention, a week after the intervention and a month after the intervention
  is a self-report measure of the impact of MS on the individual´s walking ability. Each item is scored from 1 (no limitation) to 5 (extreme limitation), with a total score ranging from 12 to 60, where higher values show higher impairment
  . MSWS-12 scale shows properties which make it suitable for use in clinical practice, concretely for patients with medium-to-high levels of walking disability
Change in The Time up and go test (TUG) | inmediatly before intervention, inmediatly after intervention, a week after the intervention and a month after the intervention
  was designed initially to measure the probability for falls among older adults, but has been validated also for other populations such as MS. For this test, the participants sit in a chair with their backs supported by the back of the chair and their arms resting on the armrests. The participants are asked to get up from the chair and walk a distance of 3 me-ters, to turn on themselves (360°) and walk back to the chair and sit down again. The TUG test has demon-strated to be highly reliable and responsive in the assessment of respectively the walking capacity and general mobility of patients with MS with mild disability
Change in The Multiple Sclerosis International QoL (Musiqol-54) | inmediatly before intervention and a month after the intervention
  This is a specific quality of life questionnaire for MS. This is a self-assessment question-naire composed of 54 items, divided in a physical and mental domain. The range goes from 0 to 100, where 100 is the highest degree of quality of life. The Spanish version of the MSQoL 54 instrument has shown to be a valid and reliable instrument for measuring qual-ity of life in patients with MS
Change in analog scale of quality of life | inmediatly beforeintervention, a week after intervention and a month after intervention
  analog scale of quality of life from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: ALBERTO JAVIER, PT, MSc, Principal Investigator — Hospital Universitario de Canarias
Locations (1):
- Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife, Spain